CLINICAL TRIAL: NCT00360503
Title: Antimicrobial Resistance in Sputum Obtained From Patients With Cystic Fibrosis (CF)
Brief Title: Antimicrobial Resistance in Cystic Fibrosis (CF)
Status: Completed | Type: Observational
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Jane L. Burns, MD, Seattle Children's Research Institute
Other Study IDs: BURNS04A0
Record Dates: First submitted 2006-08-02; First posted 2006-08-04 (Estimated); Last update posted 2009-02-10 (Estimated); Status verified 2009-02

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Antibiotic resistance; Microbiology
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bacterial isolates
Oversight: Data Monitoring Committee: No

SUMMARY:
People with cystic fibrosis (CF) often develop chronic pulmonary infections which are caused by a variety of organisms, the most predominant being Pseudomonas aeruginosa. Antibiotics are important in managing CF lung infections. Antibiotic use in CF was altered about ten years ago with the approval of inhaled tobramycin, an aminoglycoside which is effective in treating P. aeruginosa. A decade later, CF clinicians are increasingly concerned about the likelihood of induction of aminoglycoside-resistance with prolonged use of inhaled tobramycin to treat chronic P. aeruginosa airway infections. The goal of this study is to examine the current microbiology and susceptibility of organisms from CF sputum, correlate it with antibiotic use, and compare it with previous data.

DETAILED DESCRIPTION:
Aminoglycosides are one of the mainstays of antibiotic therapy in CF. They are administered parenterally in synergistic combinations with β-lactam antibiotics for acute exacerbations and used by inhalation as single agents for chronic maintenance therapy. It is well known in CF and other chronic infections that chronic use of antibiotics results in resistance. Thus, the increasing use of aminoglycosides could have dramatically changed the microbiological epidemiology of CF, since it was last examined a decade ago. It will be important to determine the current prevalence of antibiotic resistance in CF pathogens. Current antimicrobial strategies may also be contributing to the increased rate of isolation of novel and difficult to treat organisms, including intrinsically antibiotic-resistant bacteria. These issues are important both for CF clinicians and for researchers developing new antimicrobials to be used in CF.

To determine if the prevalence of P. aeruginosa resistance and the prevalence of other CF pathogens has changed over the past ten years, this multi-center cross-sectional study will enroll a contemporary cohort of patients with CF and will compare their sputum microbiology and susceptibility data with corresponding baseline data from an historical cohort consisting of patients enrolled in the prior phase 3 trials of inhaled tobramycin, conducted by PathoGenesis Corporation. (A Phase III Placebo Controlled Clinical Trial (PC-TNDS-002) to Study the Safety and Efficacy of Tobramycin in Inhalation in Patients with Cystic Fibrosis). The data set from the phase 3 trials which will be used for this research project will be anonymous.

This current study will be coordinated by the CF research team at CHRMC and aims to enroll 520 patients at approximately 50 participating sites across the United States. The contemporary cohort will include patients with CF who are ages 6 years and older and able to expectorate sputum. Patients will be enrolled from many of the same CF centers that participated in the phase 3 trials of inhaled tobramycin, and eligibility criteria will be similar to those used in the phase 3 trials. Subjects enrolled in the contemporary cohort will have a single study visit to obtain a sputum sample that will be sent to a central laboratory for culture and susceptibility testing.

ELIGIBILITY:
Inclusion Criteria:

* > 6 years of age.
* Documented sweat chloride greater than 60 mEq/mL by quantitative pilocarpine iontophoresis test or homozygous for deltaF508 genetic mutation (or heterozygous for two well-characterized mutations) and one or more clinical features consistent with CF.
* Most recent FEV1 between 25% and 75% predicted when clinically stable; must be obtained at or within 3 months prior to study visit.
* P. aeruginosa present in the most recent sputum or throat culture obtained within 6 months prior to study visit.
* Able to expectorate sputum on a routine basis.
* Written informed consent provided.

Exclusion Criteria:

* Administration of any anti-pseudomonal antibiotics by any route within 14 days prior to study visit.
* Participation in a research protocol that potentially involves antibiotic treatment within 14 days prior to study visit.
* Requiring treatment with intravenous or inhaled anti-pseudomonal antibiotics at study visit.
* B. cepacia complex present in the most recent sputum or throat culture obtained within 6 months prior to study visit.
* Post lung transplantation.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and young adults with cystic fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2006-03; Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane L Burns, MD, Principal Investigator — University of Washington and Children's Hospital and Regional Medical Center
Locations (1):
- Children's Hospital and Regional Medical Center, Seattle, Washington, United States

REFERENCES:
- [Background] Burns JL, Emerson J, Stapp JR, Yim DL, Krzewinski J, Louden L, Ramsey BW, Clausen CR. Microbiology of sputum from patients at cystic fibrosis centers in the United States. Clin Infect Dis. 1998 Jul;27(1):158-63. doi: 10.1086/514631. PMID 9675470